CLINICAL TRIAL: NCT01888614
Title: Exhaled Carbon Monoxide as a Marker of Hemolysis in Sickle Cell Disease- an Exploratory Study
Status: Withdrawn | Type: Observational
Why Stopped: Unable to secure equipment to proceed
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Jane Little, Professor, University Hospitals Cleveland Medical Center
Other Study IDs: 03-12-41
Record Dates: First submitted 2013-06-19; First posted 2013-06-28 (Estimated); Last update posted 2016-12-23 (Estimated); Status verified 2016-12

CONDITIONS: Sickle Cell Disease
Keywords: carbon mono oxide; sickle cell; hemolysis
MeSH Terms: conditions — Anemia, Sickle Cell; Hemolysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Sickle Cell Patients: Patients with Sickle Cell, over 18 years of age

SUMMARY:
The investigators propose to evaluate etCO in patients with HbSS, HbSC, and HbS-beta thalassemia during routine clinic visits, and longitudinally. Our goal is to know whether etCO differs amongst subjects with different sickle cell syndrome genotypes, and whether it is a stable marker of hemolytic rate, as reflected in routine labs obtained for clinical care (including total hemoglobin, reticulocyte count, lactate dehydrogenase, and, when sampled, total and direct bilirubin). We hope to establish whether this inexpensive and non-invasive test faithfully reflects hemolytic parameters in sickle cell syndromes.

DETAILED DESCRIPTION:
This is an observational study of sickle cell patients with the aim to measure exhaled carbon monoxide levels and to correlate with genotype and standard clinical markers of hemolysis.

Upon enrollment and at each subsequent visit, if acceptable to the patient, each subject will undergo measurement of exhaled carbon monoxide utilizing a hand held carbon monoxide monitor, MicroCO/Smoke check. Subsequent evaluations may be obtained during a routine visit, while hospitalized for a vasocclusive crises (VOC) episode, or when evaluated in the acute care clinic.

The principal study objective is to assess if exhaled carbon monoxide levels are a non-invasive marker of hemolysis in subjects with sickle cell disease (SCD).

The secondary study objective is to assess exhaled carbon monoxide levels serially in subjects with SCD, relative to vasocclusive crises, transfusion requirements, and pain syndromes.

The one inclusion criteria is for all adult sickle patients presenting for follow up at the outpatient sickle cell clinic who are capable of following simple instructions.

The exclusion criteria are a recent (2 week) history of lung infection, asthma, acute chest syndrome, or COPD exacerbation and/or a significant pulmonary dysfunction in the recent (3-6 month) past.

ELIGIBILITY:
Inclusion Criteria:

All adult sickle patients presenting for follow up at the outpatient sickle cell clinic who are capable of following simple instructions.

Exclusion Criteria:

A recent (2 week) history of lung infection, asthma, acute chest syndrome, or COPD exacerbation and/or a significant pulmonary dysfunction in the recent (3-6 month) past.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult sickle cell patients from hematology clinics at UHCMC Seidman Cancer Center would be recruited for serial measurements of exhaled CO levels, at baseline and during painful vaso-occlusive (VOC) episodes.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-06; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Exhaled Carbon Monoxide Level and hemolysis markers | Participants will be followed for the duration of two years, at baseline clinically, or while hospitalized for a VOC episode, or when evaluated in the acute care clinic for pain or symptom exacerbation.
  Exhaled Carbon Monoxide Levels will be measured serially, at clinical baseline and with symptom exacerbation.

CONTACTS AND LOCATIONS:
Overall Officials: Jane Little, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- Seidman Cancer Center, University Hospitals, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No